CLINICAL TRIAL: NCT02578771
Title: Pilot Clinical Evaluation to Characterize the in Vivo Effects of Topically Applied ZuraPrep and ZuraPrep Vehicle
Brief Title: Pilot Clinical Evaluation to Characterize in Vivo Effects of Topically Applied ZuraPrep & ZuraPrep Vehicle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zurex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ZX-ZP-0068 (MBT#865-104)
Record Dates: First submitted 2015-10-08; First posted 2015-10-19 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — citrate, isopropyl alcohol, methylene blue, parabens drug combination; Chromogranins; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ZuraPrep with 70% Isopropyl alcohol (Experimental): Test Article ZuraPrep with 70% isopropyl alcohol (IPA) will be compared with reference positive control Chloraprep
  Interventions: Drug: ZuraPrep with 70% IPA; Drug: ChloraPrep CHG/IPA Teal Tint
- ZuraPrep without 70% IPA (Experimental): Vehicle test article ZuraPrep without isopropyl alcohol will be compared with normal saline
  Interventions: Drug: ZuraPrep without 70% IPA; Other: Normal Saline
- ChloraPrep Teal Tint (Active Comparator): Test Article ZuraPrep with 70% isopropyl alcohol will be compared with reference positive control ChloraPrep [Chlorhexidine gluconate(CHG)/IPA] Teal Tint
  Interventions: Drug: ZuraPrep with 70% IPA; Drug: ChloraPrep CHG/IPA Teal Tint
- Normal Saline 0.85% (Placebo Comparator): Vehicle test article ZuraPrep without isopropyl alcohol will be compared with normal saline 0.85%
  Interventions: Drug: ZuraPrep without 70% IPA; Other: Normal Saline

INTERVENTIONS:
Drug: ZuraPrep with 70% IPA — Apply topically
  Other Names: 70% IPA
  Arms: ChloraPrep Teal Tint; ZuraPrep with 70% Isopropyl alcohol
Drug: ZuraPrep without 70% IPA — Apply topically. 0% IPA
  Other Names: ZuraPrep Vehicle
  Arms: Normal Saline 0.85%; ZuraPrep without 70% IPA
Drug: ChloraPrep CHG/IPA Teal Tint — Apply topically
  Other Names: CHG 2% / IPA 70%
  Arms: ChloraPrep Teal Tint; ZuraPrep with 70% Isopropyl alcohol
Other: Normal Saline — Apply topically
  Other Names: 0.85% Sodium Chloride (NaCl)
  Arms: Normal Saline 0.85%; ZuraPrep without 70% IPA

SUMMARY:
ZuraPrep is being evaluated for efficacy as a preoperative skin preparation solution to demonstrate its immediate and persistent antimicrobial properties. At least 72 subjects will be randomized utilizing bilateral applications on abdomen and groin. ZuraPrep active product and reference positive control will be compared; ZuraPrep non-active and negative control will be compared. Each subject will receive two of the planned treatments, one on the left side of body and one of the right. Study duration for subjects - 3 to 4 weeks.

DETAILED DESCRIPTION:
The single investigational test article, ZuraPrep solution is being evaluated for efficacy as a preoperative skin preparation solution to demonstrate its immediate and persistent antimicrobial properties. At least 72 subjects will be randomized utilizing bilateral applications on abdomen and groin.

The primary objective of this study is to characterize the in vivo effects of the ZuraPrep test article compared to the positive reference control ChloraPrep, as well as to evaluate the ZuraPrep test vehicle to the negative control, Saline, using the newly proposed sampling intervals.

This is a randomized, paired-comparisons design where each subject will receive two of the planned treatments, one on the left side of body and one on the right. Treatments will be evaluated at 30 seconds, 10 minutes and 6 hour sampling intervals compared to baseline. Status will be calculated separately for the abdomen and groin for each side of the body.

Study duration for subjects - 3 to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 18 years of age or older.
* Are in good general health.
* Have skin within 6 inches of the test sites that is free of tattoos, dermatoses, abrasions, cuts, lesions or other skin disorders.
* Cooperative and willing to follow Subject Instructions.
* Cooperative and willing to sign Consent Form and HIPAA Authorization Form.
* Have acceptable Screening Day baseline counts (CFU/cm2).

Exclusion Criteria:

* Topical or systemic antimicrobial exposure within 14 days prior to Screening Day. Restrictions include, but are not limited to antimicrobial soaps, antiperspirants/deodorants, shampoos, lotions, perfumes, after shaves, colognes, and topical or systemic antibiotics.
* Swimming in chemically treated pools or bathing in hot tubs, spas and whirlpools within 14 days prior to Screening Day.
* Use of tanning beds, hot waxes, or depilatories, including shaving (in the applicable test areas) within 14 days prior to Screening Day.
* Contact with solvents, acids, bases, fabric softener-treated clothing or other household chemicals in the applicable test areas within 14 days prior to Screening Day.
* Subjects who have a history of sensitivity to natural rubber latex, adhesive skin products (e.g., Band-Aids, medical tapes), isopropyl alcohol, citric acid, methylene blue, methylparaben, propylparaben, or chlorhexidine gluconate products.
* Subjects who have a history of skin allergies.
* Subjects who have a history of skin cancer within 6 inches of the applicable test areas.
* Subjects who are pregnant, attempting pregnancy or nursing. For all females of child-bearing potential (<60 years of age), a urine pregnancy test will be performed prior to treatment on Treatment Day.
* Subjects who have showered or bathed within 72 hours of the Screening Day or Treatment Day (sponge baths may be taken, however, the lower abdomen and upper thigh region must be avoided).
* Subjects who receive an irritation score of 1 for any individual skin condition prior to Screening Day baseline or Treatment Day baseline sample collection.
* Participation in another clinical trial in the 30 days prior to Test Day of this study (treatment with test materials in this study), or be currently enrolled in another clinical trial, or has previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Reduction of skin flora measured by Tentative Final Monograph (TFM) Proposed Amendment | 30 seconds
  calculated as log-10 CFU responder rates from baseline
Reduction of skin flora measured by 1994 TFM | 10 minutes
  calculated as log-10 CFU reductions from baseline

SECONDARY OUTCOMES:
Skin flora measurement | 6 hours
  The bacterial counts should not exceed baseline at the 6 hour sampling time

CONTACTS AND LOCATIONS:
Overall Officials: M. Hamid Barshir, MD, Principal Investigator — MicroBioTest
Locations (1):
- MicroBioTest, Sterling, Virginia, United States